CLINICAL TRIAL: NCT00772993
Title: Efficacy of RNFL / Retinal Thickness Ratio by Cirrus OCT Utilizing Spectral -Domain Technology as a Diagnostic Predictor of Glaucoma
Brief Title: Efficacy of Retinal Nerve Fiber Layer (RNFL) / Retinal Thickness Ratio by Cirrus OCT Utilizing Spectral -Domain Technology as a Diagnostic Predictor of Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Kim Chan Yun, Institute of Vision Research, Department of Ophthalmology, Yonsei University School of Medicine, Severance Hospital.
Other Study IDs: 4-2008-0340
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Glaucoma; Myopia
Keywords: glaucoma; myopia; myopia with glaucoma; normal control
MeSH Terms: conditions — Glaucoma; Myopia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Primary open angle glaucoma
- 2: Normal Control
- 3: Myopia with no evidence of glaucoma
- 4: Myopia with evidence og glaucoma

SUMMARY:
Glaucoma is presumed to be an axonal disease which starts at the lamina cribrosa. This assumption has led to the monitoring of the retinal nerve fiber layer thickness for the diagnosis and monitoring of progression of glaucoma. However, varying disc size, myopia and tilted discs affect the thickness of the retinal nerve fiber layer. This study aims to ascertain the ration of the retinal nerve fiber layer against full retina as a predictor of glaucoma diagnosis and progression.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma
* Myopia
* Myopia with evidence of glaucoma
* Normal controls

Exclusion Criteria:

* Evidence of retinal disease
* BCVA < 0.4
* Secondary glaucoma due to intraocular inflammation
* Lens induced glaucoma
* Tumor induced glaucoma
* Neovascular glaucoma

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: prospective consecutive recruitment from a tertialry glaucoma subspecialty practise
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Ratio of RNFL / Full thickness retina | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Severance Hospital, Yonsei University School of Medicine, Seoul, South Korea